CLINICAL TRIAL: NCT06329336
Title: Parenting Support for Justice Involved Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Liliana Lengua, Professor: Psychology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019653; UL1TR002319 (NIH)
Record Dates: First submitted 2024-03-08; First posted 2024-03-25 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Parenting; Well-Being, Psychological; Mental Health Wellness 1
Keywords: parenting intervention; mindfulness; well-being; re-entry
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preventive Behavioral Parenting Program (Experimental): This preventive parenting intervention combines behavioral parenting and mindfulness-based well-being practices to support effective parenting.
  Interventions: Behavioral: Social Emotional Competence for Children and Parents

INTERVENTIONS:
Behavioral: Social Emotional Competence for Children and Parents — This preventive parenting intervention combines behavioral parenting and mindfulness-based well-being practices to support effective parenting.

SUMMARY:
Together with the Community Care Team of King County Community Partnership for Transition Solutions (KCCPTS), the investigators propose to collaborate in adapting parenting intervention(s) to support the well-being and effective parenting of parents re-entering the community, as well as that of their children's primary caregiver. The aim is promoting the well-being of the parents/caregivers and their children, fostering positive child development, and ultimately, preventing the intergenerational transmission of adversity. The KCCPTS Community Care Team includes re-entry navigators who have lived experience of adversity and incarceration, bringing their unique insights regarding the re-entry experience, from both personal and professional experiences. This study will evaluate a task-sharing approach to offering formerly incarcerated parents and their families a parenting support intervention. That is, re-entry navigators will be trained to deliver evidence-based parenting interventions. This increases the feasibility and accessibility of the program, particularly because facilitators have shared experiences and trusted connections with their clients. This project proposes four main activities: 1) conduct focus groups with parents re-entering the community to better understand their parenting needs, 2) work with KCCPTS re-entry navigators to incorporate information from their experience and the focus group to adapt a parenting intervention, 3) train re-entry navigators to deliver the program, and 4) conduct a preliminary evaluation of the impact of the program on parents' well-being and parenting when the program is delivered by KCCPTS re-entry navigators. If this preliminary evaluation shows promise in supporting parent well-being and parenting effectiveness, the investigators will seek funding to conduct a larger, more rigorous evaluation.

DETAILED DESCRIPTION:
Research Plan: The incarceration of a parent is associated with a higher likelihood of children living in poverty, increased likelihood of needing mental health services and involvement in child protective service, increases in teen crime, and significant decreases in educational attainment and adult employment. Incarceration disproportionately affects families of color and those living in poverty, and impacts children's long-term ability to emerge from poverty in adulthood, increasing the rate of intergenerational transmission of adversity and incarceration. Thus, it is critical to support families experiencing the incarceration of a parent. It is equally important to provide parents returning home from prison with programs that equip them with parenting strategies and techniques to buffer the potentially adverse outcomes of parental incarceration on their children's socioemotional development. It may be the case that parenting programs post release may in fact serve to reduce recidivism.

The proposed project arises out of a request from KCCPTS, stemming from their recognition of the parenting needs of their clients and the desire to break the cycle of intergenerational transmission of adversity and incarceration. Parents returning to their families after incarceration have unique experiences and needs as they work to strengthen their relationships with their children. In addition to potential challenges connecting with and parenting their children, they often experience mental health issues related to their adverse childhood experiences (ACEs) and incarceration. This may contribute to the intergenerational transmission of adversity and incarceration. While parenting interventions exist, they do not specifically address the unique needs of formerly incarcerated parents. Additionally, they are expensive or hard to access, and do not explicitly address the mental and emotional well-being of the parent to support more effective parenting. Caregivers for the children while the parent was incarcerated, usually the other parent or a grandparent, also experience adversity and challenges with parenting, and may benefit from support as they surrender the parenting role or co-parent with the formerly incarcerated parent. The proposed project would equip staff with tools to more effectively support the well-being of parents, children and caregivers through a task-sharing approach.

A task-sharing model for prevention is a promising approach to addressing the need for interventions in low-resource settings with a limited workforce to meet the need. In task-sharing, staff currently working with community organizations serving children and families are trained to deliver prevention programs. These staff often have developed trusting relationships with the families they serve, and thus interventions can be incorporated into regular services at little additional cost to the organization. Finally, after staff are trained, the tools and resources remain with the community. Such an approach holds tremendous promise for making preventive parenting interventions more accessible in communities that often do not have access to evidence-based interventions due to resource, language, or time barriers. Research evaluating such approaches provides knowledge about innovative ways to improve mental health in low-resource communities, and a task-sharing approach, if shown to be effective, offers a generalizable and scalable approach to improving community mental health over time.

Project Aims: The investigators aim to evaluate a task-sharing approach to offering formerly incarcerated parents and their families a parenting support intervention. That is, re-entry navigators will be trained to deliver evidence-based behavioral parenting intervention(s) that promote children's social-emotional and behavioral well-being. This will include cognitive-behavioral and mindfulness practices for supporting parent well-being. The task-sharing approach increases the feasibility and accessibility of the program, particularly because facilitators have shared experiences and trusted connections with their clients. This project proposes four main activities: 1) conduct focus groups with parents re-entering the community to better understand their parenting needs and challenges, 2) work with KCCPTS re-entry navigators to incorporate information from their experience and the focus group to adapt an existing parenting intervention, 3) train re-entry navigators to deliver the program, and 4) conduct a preliminary evaluation of the impact of the program on parents' well-being and parenting when the program is delivered by KCCPTS re-entry navigators.

Research Plan: Preliminary studies. The Center for Child and Family Well-being (CCFW) has convened a multidisciplinary group of collaborators to conduct research on supporting families experiencing the incarceration of a parent. The goal is to evaluate approaches to supporting the whole family experiencing a parent's incarceration. Collectively, the researchers have developed and implemented interventions for parents who are currently or formerly incarcerated (Charles, Pace) as well as a parenting program for parents living in poverty or who are experiencing homelessness (Lengua). The proposed study would add to this body of evidence that a task-sharing approach can address accessibility and feasibility of prevention programs.

Research design. This project includes 4 research phases related to the study aims:

Aim 1: Conduct 2 focus groups with parents re-entering the community to better understand their parenting needs. KCCPTS will facilitate the invitation of 5-7 women and 5-7 men who are parents re-entering the community to participate in 2 separate focus groups led by a UW research coordinator. The goal of the focus group is to obtain information on parents' perspectives on their experiences, goals, and preferred approaches to supporting their relationships with their children. Focus groups will be 1.5 hours and held at KCCPTS facilities. Structured questions with potential follow-up discussion questions will be developed together with KCCPTS staff and clients.

Aim 2: Work with KCCPTS re-entry navigators and clients to incorporate their experiences and focus group information to adapt an existing parenting intervention to be more relevant to formerly incarcerated individuals. Re-entry navigators' and parents' expertise will be used to select and adapt a program (e.g., Parenting Inside Out [PIO, Eddy et al., 2008]; Pathways for Parents [P4P, Charles et al., in press]; Social, Emotional Attunement for Children & Parents [SEACAP, Lengua et al., 2018]). KCCPTS and research team members will incorporate changes to the selected program(s) based on focus group findings and staff experiences. Changes will be incorporated into program manuals to standardize delivery.

Aim 3: Train re-entry navigators to deliver the program. KCCPTS staff who have already participated in the REAL Pro training will participate in 8-10 hours of training in the concepts and practices of behavioral parenting and delivering parenting, cognitive-behavioral, and mindfulness content. Training will be delivered by Dr. Charles (for PIO/P4P), Dr. Lengua (SEACAP), and CCFW staff.

Aim 4: Conduct a preliminary evaluation of intervention effects on parents' and children's well-being and parenting behaviors when the program is delivered by KCCPTS re-entry navigators. Navigators will offer 2 groups, one each to mothers and fathers, with 6-8 participants in each group. The evaluation will include pre-/posttest assessments conducted by RAs. Assessments will include measures of participant and child mental health, well-being, parenting behaviors and sense of competence, and satisfaction ratings. Assessments will be approximately 30 minutes, including obtaining informed consent and administering all measures.

Measures. Assessments will include CCFW's program evaluation protocol: demographics, depression (PHQ-9), anxiety (GAD7), Difficulties with Emotion Regulation, Self-Compassion Scale, Brief Resilience Scale, Flourishing Scale, stress (General Life Events and Perceived Stress Scales), ACEs, Everyday Discrimination Scale, Positive Relations with Others subscale of the Psychological Well-being measure, Parenting Behavior Inventory - Very Short Form, Parent Sense of Confidence Scale, Strengths and Difficulties Questionnaire of child social-emotional and behavioral adjustment.

Impact: Evidence from the proposed study will be shared with KCCPTS in planning ongoing collaboration, as well as in international conference presentations. The findings would support a more rigorous evaluation of the effectiveness of preventive interventions when delivered by staff working in community organizations serving families experiencing adversity. With adequate funding, future research can explore the critical downstream impact, including improved developmental outcomes for children and decreases in the need for more intensive mental health services for parents. Evaluation of a scalable model for delivering parenting interventions to promote well-being in parents and children offers a promising approach to addressing social inequities by ensuring access to evidence-based prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* Formerly Incarcerated
* Parent with child between the ages of 2 and 12 years

Exclusion Criteria:

* Does not have reasonable proficiency in English
* Diagnosed cognitive disability that would limit ability to complete assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Parenting Behavior Inventory - Very short Form | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring parental warmth and consistency, scores range from 0 to 4, high scores reflect higher warmth and consistency.
PHQ-9 Depressive Symptoms | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring mental health - Depressive symptoms, scores range from 0 to 27, higher scores indicate a greater number or severity of depressive symptoms
GAD-7 Anxiety Symptoms | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring mental health - Anxiety Symptoms, scores range from 0 to 21, higher scores indicated a greater number of severity of anxiety symptoms
Brief Resilience Scale | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring well-being - Resilience, scores range from 6 to 30, higher scores indicating greater resilience
Self-Compassion Scale - Short Form | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring well-being - mindfulness and self-compassion, scores range from 12 to 60, higher scores indicate greater self-compassion.
Strengths and Difficulties Questionnaire | From enrollment to the end of treatment at 6 weeks
  Questionnaire measuring child social-emotional and behavioral adjustment, scores range from 0 to 50, higher scores indicate great emotional and behavioral difficulties